CLINICAL TRIAL: NCT03829111
Title: Pilot Study to Evaluate the Biologic Effect of CBM588 in Combination With Nivolumab/Ipilimumab for Patients With Metastatic Renal Cell Carcinoma
Brief Title: CBM588, Nivolumab, and Ipilimumab in Treating Patients With Stage IV or Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18523; NCI-2019-00248 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18523 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Advanced Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (nivolumab, ipilimumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 5, patients receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab
- Arm II (CBM588, nivolumab, ipilimumab) (Experimental): Patients receive clostridium butyricum CBM 588 probiotic strain PO BID, nivolumab IV over 30 minutes on day 1, and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 5, treatment with clostridium butyricum CBM 588 probiotic strain and nivolumab repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Clostridium butyricum CBM 588 Probiotic Strain; Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Drug: Clostridium butyricum CBM 588 Probiotic Strain — Given PO
  Other Names: C. butyricum CBM 588 Probiotic Strain; C. butyricum MIYAIRI Strain; C. butyricum Strain MIYAIRI 588; CBM 588; CBM588; Clostridium butyricum MIYAIRI 588; Clostridium butyricum MIYAIRI 588 Probiotic Strain; MIYAIRI 588; MIYAIRI 588 Strain of C. butyricum
  Arms: Arm II (CBM588, nivolumab, ipilimumab)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase I trial studies how well CBM588 works when given together with nivolumab and ipilimumab in treating patients with kidney cancer that is stage IV or has spread to other places in the body (advanced). CBM588 is a probiotic that may help to increase the effect of immunotherapy. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving CBM588, nivolumab, and ipilimumab may work better in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of clostridium butyricum CBM 588 probiotic strain (CBM588) (in combination with nivolumab/ipilimumab) on the gut microbiome in patients with metastatic renal cell carcinoma (mRCC).

SECONDARY OBJECTIVES:

I. To evaluate the effect of CBM588 on the clinical efficacy of the nivolumab/ipilimumab combination.

II. To assess the effect of CBM588 on systemic immunomodulation of the nivolumab/ipilimumab combination in patients with mRCC.

III. To assess the effect of CBM588 on toxicities such as diarrhea and nausea using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 criteria with the nivolumab/ipilimumab combination in patients with mRCC.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 5, patients receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive clostridium butyricum CBM 588 probiotic strain orally (PO) twice daily (BID), nivolumab IV over 30 minutes on day 1, and ipilimumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 5, treatment with clostridium butyricum CBM 588 probiotic strain and nivolumab repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide informed consent for the trial
* Histological confirmation of RCC with a clear-cell component
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (American Joint Committee on Cancer [AJCC] stage IV) RCC
* Intermediate or poor risk disease by International Metastatic RCC Database Consortium (IMDC) classification
* No prior systemic therapy for RCC with the following exception:

  * One prior adjuvant or neoadjuvant therapy for completely resectable RCC if such therapy did not include an agent that targets PD-1 or PD-L1 and if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Any ethnicity or race
* Calculated creatinine clearance >= 30 milliliters per minute (mL/min) per the Cockcroft and Gault formula or serum creatinine < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN if liver metastases are present)
* Total bilirubin < 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin up to 3.0 mg/dL)
* White blood cells (WBC) > 2,000/mm^3
* Neutrophils > 1,500/mm^3
* Platelets > 100,000/mm^3

Exclusion Criteria:

* Presence of untreated brain metastases. Patients with treated brain metastases must be stable for 4 weeks after completion of treatment and have documented stability on pre-study imaging. Patients must have no clinical symptoms from brain metastases and have no requirement for systemic corticosteroids amounting to > 10 mg/day of prednisone or its equivalent for at least 2 weeks prior to first dose of study drug. Patients with known leptomeningeal metastases are excluded, even if treated

  * Not recovered to =< grade 1 toxicities related to any prior therapy before administration of study drug
* Favorable risk disease by IMDC classification
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo or type I diabetes mellitus or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll
* Active interstitial lung disease (ILD)/pneumonitis or history of ILD/pneumonitis requiring treatment with systemic steroids
* Baseline pulse oximetry less than 92% "on room air"
* Current use, or intent to use, probiotics, yogurt or bacterial fortified foods during the period of treatment
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Uncontrolled adrenal insufficiency
* Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
* Not recovered to =< grade 1 toxicities related to any prior therapy before administration of study drug
* Women who are pregnant or breastfeeding
* History of myocarditis or congestive heart failure (as defined by New York Heart Association functional classification III or IV), as well as unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction 6 months prior to study entry
* White blood cells (WBC) < 2,000/mm^3
* Neutrophils < 1,500/mm^3
* Platelets < 100,000/mm^3
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN) (> 5 x ULN if liver metastases are present)
* Total bilirubin > 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin 3.0 mg/dL)
* Calculated creatinine clearance < 30 millimeters per minute (mL/min) per the Cockcroft and Gault formula or serum creatinine > 1.5 x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Change in Bifidobacterium composition of stool | Baseline up to week 12
  Will be assessed for patients on both arms.

SECONDARY OUTCOMES:
Change in Shannon index | Baseline up to week 12
  Using translational methods, will compute the Shannon index at baseline for a comparison of microbial diversity.
Best overall response | Up to 2 years
  Will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST). The association between treatment arm and overall response as per RECIST criteria (response observed versus [vs] not observed) will be examined using Fisher's exact test.
Progression-free survival (PFS) | From enrollment to progression, assessed up to 2 years
  The difference in progression free survival across the two groups will be explored graphically using Kaplan-Meier survival plots. Median PFS time for each of the two arms will be reported and Cox proportional hazards model will be used to estimate the hazard ratio and its confidence interval.

OTHER OUTCOMES:
Change in proportion of circulating regulatory T-cells (Tregs) | Baseline up to 2 years
  Using translational methods will estimate the proportion of Tregs in the blood. This will be assessed graphically across serial timepoints of blood collection to ascertain any trends. Will compare the proportion of circulating Tregs with nivolumab/ipilimumab alone versus nivolumab/ipilimumab with clostridium butyricum CBM 588 probiotic strain (CBM588).
Change in proportion of circulating myeloid-derived suppressor cells (MDSCs) | Baseline up to 2 years
  Using translational methods will estimate the proportion of MDSCs in the blood. This will be assessed graphically across serial timepoints of blood collection to ascertain any trends. Will compare the proportion of circulating MDSCs with nivolumab/ipilimumab alone versus nivolumab/ipilimumab with CBM588.
Change in IL-6, IL-8, and other cytokines/chemokines levels | Baseline up to 2 years
  Using translational methods will estimate the proportion of serum cytokines in the blood. This will be assessed graphically across serial timepoints of blood collection to ascertain any trends. Will compare the IL-6, IL-8, and other cytokines/chemokines with nivolumab/ipilimumab alone versus nivolumab/ipilimumab with CBM588.
Change in toxicities | Baseline up to 2 years
  Will compare toxicities, such as diarrhea and nausea, using Common Terminology Criteria for Adverse Events version 5 with nivolumab/ipilimumab alone versus nivolumab/ipilimumab with CBM588.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta K Pal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Villemin C, Six A, Neville BA, Lawley TD, Robinson MJ, Bakdash G. The heightened importance of the microbiome in cancer immunotherapy. Trends Immunol. 2023 Jan;44(1):44-59. doi: 10.1016/j.it.2022.11.002. Epub 2022 Dec 1. PMID 36464584
- [Derived] Dizman N, Meza L, Bergerot P, Alcantara M, Dorff T, Lyou Y, Frankel P, Cui Y, Mira V, Llamas M, Hsu J, Zengin Z, Salgia N, Salgia S, Malhotra J, Chawla N, Chehrazi-Raffle A, Muddasani R, Gillece J, Reining L, Trent J, Takahashi M, Oka K, Higashi S, Kortylewski M, Highlander SK, Pal SK. Nivolumab plus ipilimumab with or without live bacterial supplementation in metastatic renal cell carcinoma: a randomized phase 1 trial. Nat Med. 2022 Apr;28(4):704-712. doi: 10.1038/s41591-022-01694-6. Epub 2022 Feb 28. PMID 35228755